CLINICAL TRIAL: NCT07057518
Title: The Effect of Emotional Freedom Technique on Psychological Health and Well-being in People With Type 2 Diabetes.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 642-642-11
Record Dates: First submitted 2025-07-07; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Emotional Freedom Technique; RCTs
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: People with Type 2 diabetes who meet the inclusion criteria for the research will use the Random.org website to allocate participants to the Emotional Freedom Technique and Control group.
Who Masked: Outcomes Assessor
Masking Description: The analysis of the research will be done by the other researcher, not by the researcher who applied it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional freedom technique group (Experimental): The EFT application will be implemented by the researcher who has been trained in this subject, in the most quiet and calm environment possible, in a position where the individuals are comfortable. There are basic steps to be followed in EFT application. Thought Field Therapy (TFT), developed by Callahan, based on Craig, uses different click points for specific psychological conditions, while EFT has 12 energy click points in the same specified order to treat every emotional problem, It is called 'Basic Recipe'
  Interventions: Behavioral: emotional freedom technique
- Control group (No Intervention): No intervention was made to the people with Type 2 diabetes in the control group.

INTERVENTIONS:
Behavioral: emotional freedom technique — The EFT application will be implemented by the researcher who has been trained in this subject, in the most quiet and calm environment possible, in a position where the individuals are comfortable. There are basic steps to be followed in EFT application. Thought Field Therapy (TFT), developed by Callahan, based on Craig, uses different click points for specific psychological conditions, while EFT has 12 energy click points in the same specified order to treat every emotional problem, It is called 'Basic Recipe'
  Arms: Emotional freedom technique group

SUMMARY:
Type 2 diabetes is a major meatbolic condition. People living with Type 2 diabetes come across a wide range of health issues, including psychological health. Specifically, diabetes distress are in high levels among them. Diabetes distress is associated with psychological states such as anxiety, lower levels of self-care, and higher hemoglobin A1c (HbA1c) levels. The Emotional Freedom Technique consists of cognitive and somatic components and is used to heal an individual's negative emotions and manage associated emotional and physical disorders. The basic principle of this technique is to regulate the flow of energy by stimulating the meridian system and to relax the individual while focusing on the emotional reactions that lead to disability. Although the prevalence of psychological problems associated with T2DM and diabetes is increasing, there are not enough studies showing the effect of Emotional Freedom Technique on the psychological well-being of T2DM individuals.

DETAILED DESCRIPTION:
Worldwide, 589 million adults (aged 20-79) live with diabetes (IDF, 2025). This number is projected to rise to 853 million by 2050. The latest International Diabetes Federation Diabetes Atlas (2025) reports that 11.1% (or 1 in 9) of the adult population (aged 20-79) live with diabetes, and 4 in 10 are unaware that they have the condition. More than 90% of people with diabetes have type 2 diabetes (T2DM) due to socioeconomic, demographic, environmental, and genetic factors. The main factors contributing to the increase in T2DM are: urbanization, aging population, decreasing physical activity levels, and increasing prevalence of overweight and obesity. T2DM is associated with microvascular and macrovascular complications. T2DM can cause complications due to a two- to four-fold increase in impaired macrovascular circulation and a 10- to 20-fold impairment in microvascular circulation compared to people without diabetes (Gregg, 2019; Mbanya and Sobngwi, 2003). Microvascular complications, namely peripheral neuropathy, retinopathy and nephropathy, result from damage to small blood vessels in the nerves, retina and kidneys, respectively. Macrovascular complications result from damage to large vessels of the heart, brain and legs, causing heart disease (ischemic heart disease), cerebrovascular disease and peripheral vascular disease, respectively (IDF, 2022). Approximately one in three people with diabetes already has microvascular complications when diagnosed with T2DM, and the risk of developing cardiovascular complications is 2-2.5 times higher in people with diabetes compared to people without diabetes (Dal Canto, 2019). In addition, diabetes is a chronic metabolic disease that affects social and mental states, including the psychological well-being of people living with it. For example, a large-scale, cross-sectional study of the Diabetes Attitudes, Wants and Needs (DAWN) study results from around the world showed that 13.8% of 8596 DM patients in 17 countries may have depression, and approximately 50% of patients may have depression (Burns et al. 2013). Diabetes-related distress is a unique emotional problem that is directly related to the burden and anxiety felt by T2DM patients. Diabetes-related distress was found in 60.5% of T2DM patients. With this in mind, it is important to identify and support patients with physical and psychosocial problems early in the course of diabetes, as this may affect their ability to adapt or take adequate responsibility for self-care.

Diabetic distress is associated with psychological states such as anxiety, lower levels of self-care, and higher hemoglobin A1c (HbA1c) levels. Previous studies have shown that depression and anxiety are associated with an increased risk of diabetes complications (Park et al. 2024). The management of T2DM involves complex components aimed at reducing the numerous, wide-ranging complications associated with the condition. In particular, previous studies have found that psychological interventions have a significant effect on diabetic stress and anxiety levels. One of the psychological interventions in T2DM individuals is the Emotional Freedom Technique. This technique is a method derived from energy psychotherapy. The Emotional Freedom Technique consists of cognitive and somatic components and is used to improve the individual's negative emotions and manage associated emotional and physical disorders. The basic principle of this technique is to regulate the energy flow by stimulating the meridian system and to relax the individual while focusing on the emotional reactions that lead to disability. Previous meta-analyses report that this technique is one of the most recognized and widely used types of energy therapy and is effective in the management of stress as well as anxiety, depression, burnout and phobias. A systematic review and meta-analysis of randomized and non-randomized trials of the clinically applied Emotional Freedom Technique for the treatment of depression found that this technique is as effective as cognitive behavioral therapy (Nelms et al. 2016). However, although the prevalence of psychological problems associated with T2DM and diabetes is increasing, there are not enough studies showing the effect of Emotional Freedom Technique on the psychological well-being of T2DM individuals. Therefore, it is thought that this study will lead to future studies.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years of age,
* having type 2 diabetes,
* no psychiatric diagnosis
* agreeing to participate in the study.

Exclusion Criteria:

* be under 18 years of age,
* have type 1 diabetes or gestational diabetes,
* attend any course on coping with diabetes distress and anxiety,
* have advanced mental health problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
WHO-5 | Two months
  The WHO-5 scale is used to measure and evaluate an individual's emotion or happiness. The raw score is calculated by summing the five item scores and ranges from 0 to 25, with 0 representing the worst possible quality of life and 25 representing the best possible quality of life.
Diabetes Stress Scale | Two months
  The scale is used to assess diabetes distress. The diabetes stress scale demonstrates good internal consistency, indicating that the component questions measure a similar construct. Higher scores-that is, scores above 3 on the diabetes stress scale-indicate greater levels of diabetes distress and have been found to be significantly associated with suboptimal lifestyle and higher HbA1c.
General Anxiety Scale - 7 | Two months
  The scale was used to measure the severity of anxiety symptoms. Total scores range from 0 to 21, with scores of 5, 10, and 15 representing mild, moderate, and severe anxiety thresholds, respectively, and were used to create a four-category ordinal variable. A cut-off point of 10 was used to distinguish between anxiety and no anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)